CLINICAL TRIAL: NCT01604603
Title: The Clinical and Biochemical Characteristics in Women With Different Menstrual Pattern
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Ming-I Hsu, Taipei Medical University WanFang Hospital, Taipei Medical University WanFang Hospital
Other Study IDs: WFH-TMU-RetroMcLab-201203022
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Regular Menstrual Cycle; Irregular Menstrual Cycle
MeSH Terms: conditions — Menstruation Disturbances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control
- Oligomenorrhea
- Amenorrhea
- premature ovarian failure

SUMMARY:
Background: Menstrual disturbance is the major complain in reproductive age women, the clinical and biochemical characteristics of women with different menstrual disturbance had not been well-understood. Objective: To study the clinical and biochemical characteristics of women with oligomenorrhea, amenorrhea, and premature ovarian failure. Method: Retrospective study, medical records reviewed in patients who visited to outpatient clinic of Reproductive Medicine in Taipei Medical University - Wan Fang Hospital form 2009 Jan. 1 to 2011 Nov. 31. Including criteria: Patients had sufficient medical records (anthropometric, endocrine, metabolic, lipid parameters) and age less than 45. Excluding criteria: (1) Women who experienced menarche <3 years before the beginning of the study; (2) Women who received hormones or drugs for major medical diseases; (3) Women who presented ovarian cysts or ovarian tumors, uterine abnormality; (4) Women who were >45 years old.

ELIGIBILITY:
Inclusion Criteria:

* Patients had sufficient medical records (anthropometric, endocrine, metabolic, lipid parameters) and age less than 45.

Exclusion Criteria:

1. Women who experienced menarche <3 years before the beginning of the study;
2. Women who received hormones or drugs for major medical diseases;
3. Women who presented ovarian cysts or ovarian tumors, uterine abnormality;
4. Women who were >45 years old.

Ages: 13 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients had sufficient medical records (anthropometric, endocrine, metabolic, lipid parameters) and age less than 45.
Sampling Method: Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2012-04; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming I Hsu, MD, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- WanFang Medical Center at Taipei Medical University, Taipei, Taiwan, Taiwan